CLINICAL TRIAL: NCT04218175
Title: Effects of Neuromobilization on Median Nerve Elasticity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Yasemin Çırak, Physiotherapist, PhD, Associate Professor, Istinye University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 005
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Median Nerve Disease
Keywords: neuromobilization; elasticity; shear wave elastography
MeSH Terms: conditions — Median Neuropathy

STUDY DESIGN:
Intervention Model Description: The researcher who performed shear wave elastography did not know which group the case was evaluated during the measurement.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- neuromobilization stretching group (Experimental): In the neuromobilization stretching group; The subjects were brought to shoulder depression and 90 degrees of abduction while the dominant side forearms were supination. In this position, median nerve stretching was performed by extending the participant's head to the opposite side while flexing the wrist and finger. After waiting for 30 seconds in this position, the wrist and head were moved to the neutral position and the participants relaxed.
  Interventions: Other: neuromobilization exercises
- neuromobilization shifting group (Experimental): In the neuromobilization shifting group, the subjects were brought to shoulder depression and 90 degrees of abduction while the dominant forearms were supination. In this position, the participant flexed his wrist and fingers while lateral flexion of his head to the opposite side, and flexed his wrist and fingers while lateral flexion of the head to the same side. Thus, the participants performed median nerve shift.
  Interventions: Other: neuromobilization exercises
- Control Group (No Intervention): The dominant sides of the individuals are experimental sides and the other nondominant sides of the participants are control sides. And no intervention was made. All measurements were done bilaterally before and after.

INTERVENTIONS:
Other: neuromobilization exercises — Median nerve neuromobilization (stretching and shifting) was performed. For median nerve stretching; The subjects were brought to shoulder depression and 90 degrees of abduction while the dominant side forearms were supination. In this position, median nerve stretching was performed by extending the participant's head to the opposite side while flexing the wrist and finger. After waiting for 30 seconds in this position, the wrist and head were moved to the neutral position and the participants relaxed. For median nerve shift; The subjects were brought to shoulder depression and 90 degrees of abduction while the dominant side forearms were supination. In this position, the participant flexed his wrist and fingers while lateral flexion of his head to the opposite side, and flexed his wrist and fingers while lateral flexion of the head to the same side.
  Arms: neuromobilization shifting group; neuromobilization stretching group

SUMMARY:
Purpose: The aim of this study was to investigate the effect of median nerve neuromobilization on median nerve elasticity using shear wave elastography.

Methods: The study included 36 healthy volunteers (72 upper extremities) aged 18-30 years. Inclusion criteria; no known systemic neuromuscular and metabolic diseases, no nerve impingement syndrome, and no upper extremity bone-tendon-muscle surgery in the last six months. Sociodemographic data of the participants were recorded. Wrist flexion and extension bilaterally with universal goniometer and finger grip strength bilaterally were measured with pinchmeter. Median Nerve Stress Test was performed. Median nerve elasticity was measured by Shear Wave Ultrasound Elastography. The extremity of the dominant side as a study group and the non-dominant side as a control group were measured bilaterally. Median nerve neuromobilization (stretching (n = 18) and shifting (n = 18)) was applied to the upper extremities of the dominant side. The application was carried out as 3 sets in one session. Evaluations were repeated after application.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 years of age
* Healthy individuals without any known systemic disease

Exclusion Criteria:

* Those who have undergone an upper extremity bone-tendon-muscle operation in the last six months
* People with a systemic disease such as rheumatoid arthritis, diabetes mellitus
* Patients with any neuromuscular disease

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-25 (Actual)

PRIMARY OUTCOMES:
Median Nerve Tension Test | 4 weeks
  The test was performed in a position with shoulder depression and 90 degrees abduction and external rotation, elbow 90 degrees flexion, forearm full supination, and wrist and fingers fully extended. Maintaining this position, the elbow was passively extended and the tension of the median nerve was tested. The test was stopped at the point where the patient felt pain and tension, and the angle at the elbow was measured by a universal goniometer.
Median nerve elasticity with Shear Wave Ultrasound Elastography | 4 weeks
  The nerve elasticity was measured by measuring the velocity of shear waves in the median nerve by means of high frequency ultrasound waves.
Bilaterally finger grip strength with pinchmeter | 4 weeks
  finger grip strength was measured bilaterally by pinch meter.

CONTACTS AND LOCATIONS:
Locations (1):
- İstinye University, Istanbul, Turkey (Türkiye)